CLINICAL TRIAL: NCT02317926
Title: Desiccated Thyroid Extract Versus Synthetic T3/T4 Combination (ThyrolarTM) Versus L-T4 Alone in the Therapy of Primary Hypothyroidism With Special Attention to the Gene Polymorphism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mohamed K.M. Shakir, Staff Endocrinologist, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 397401-1
Record Dates: First submitted 2014-12-08; First posted 2014-12-17 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism | interventions — Thyroxine; Triiodothyronine; Thyroid (USP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Levothyroxine Plus Liothyronine Group (Active Comparator): Levothyroxine Plus Liothyronine Group
  Interventions: Drug: Levothyroxine Plus Liothyronine
- Levothyroxine Group (Active Comparator): Levothyroxine Group
  Interventions: Drug: Levothyroxine
- Desiccated Thyroid Extract Group (Active Comparator): Desiccated Thyroid Extract Group
  Interventions: Drug: Desiccated Thyroid Extract

INTERVENTIONS:
Drug: Levothyroxine
  Arms: Levothyroxine Group
Drug: Levothyroxine Plus Liothyronine
  Arms: Levothyroxine Plus Liothyronine Group
Drug: Desiccated Thyroid Extract
  Arms: Desiccated Thyroid Extract Group

SUMMARY:
The proposed study design is a prospective, randomized, double-blind, crossover study. After informed consent is obtained, patients will be randomized to receive either desiccated thyroid in capsules, or L-T4/L-T3 (ThyrolarTM) in capsules, or L-T4 alone capsules. All study participants, physician investigators, those administering the neurocognitive tests and those analyzing test results will be blinded throughout the study.

Subjects will undergo memory testing, a disease specific symptom questionnaire, a general mental health assessment, a complete physical examination, baseline EKG, and biochemical testing consisting of serum TSH, free T4, total T4, total T3, free T3, T3 resin uptake, reverse T3, sex hormone binding globulin (SHBG), serum iodine, a lipid panel, insulin, glucose and leptin. This testing and DXA scan of body composition will be performed at baseline and after each 3 month treatment period. Deiodinase type 2 (DIO2) polymorphisms analyses - will also be performed at the beginning of the study and the results will be blinded to the investigators performing the memory testing.

After 5-6 weeks on the study medication, TSH levels will be checked and the medication adjusted to maintain TSH level between 0.46-4.68 mIU/L. Once the TSH level is in the desired range, subjects will continue the medication for an additional 6 weeks. Subjects will then be crossed-over to the other treatment arm for 3 months. Again, testing will be performed after each treatment period. Finally the subjects will again switched over to the 3rd arm and testing will be performed after treatment period.

A cross-over design is preferred because we are assessing subjective symptoms such as clinical well-being and other parameters. Therefore, we will be able to evaluate the effectiveness of L-T4/T3 (ThyrolarTM) vs DTE vs T4 alone in the same patientssubjects. This is also supported by the previous study by Escobar-Morreale et al.

Additionally, the Wechsler memory scale, DEXA for body composition, measurment of reverse T3, insulin, leptin, and DIO2 polymorphisms analysis will be included for the research portion of this study. Further, the frequency of serum blood draws, for research purposes, will be at intervals of 0, 6, 12, 18, 24, 30 and 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be between the ages of 18 to 65 and will have been on levothyroxine for primary hypothyroidism for at least 6 months
* Department of Defense beneficiaries living within 60 miles of Besthesda, MD

Exclusion Criteria:

* Subjects will be excluded if they have the following problems: pregnancy, plan for pregnancy in the next 12 months, cardiac disease, especially coronary artery disease, chronic obstructive lung disease, malabsorption disorder, gastrointestinal surgeries, significant renal or liver dysfunction, seizure disorders, thyroid and non-thyroid active cancers, uncontrolled psychosis, psychotropic medication use, steroid use, amiodarone, chemotherapy for cancer, iron supplement more than 325mg per day, carafate/ proton pump inhibitor use, cholestyramine use, and those with recent orders who are expected to move out of the geographic area, age less than 18 years old or older than 65 years old. Patients scheduled for deployment will be excluded.
* Subjects with subclinical hypothyroidism will be excluded. If we include patients with subclinical hypothyroidism, it will be difficult to assess the outcomes. This is because only a very small percentage of patients with subclinical hypothyroidism benefit from thyroid hormone therapy and therefore, a cross-over study as done in this project will not show a difference between the therapies.
* Females of child-bearing age will be screened with initial assessment for pregnancy as part of standard of care (eg history of amnenorrhea and/or positive pregnancy testing via hCG). There is no experience in using desiccated thyroid extract in pregnant women and there is no published paper in this area. Desiccated thyroid extract is rated Category-A drug in pregnancy which means there are no known risks to the fetus.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2015-05; Primary Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Wechsler memory scale, fourth edition (WMS-IV) | 3 months
  Pearson, PsychCorp, San Antonio, Texas
Beck Depression Inventory | 3 months
  Pearson, PsychCorp
Thyroid Symptom Questionnaire (TSQ) | 3 months
  Clyde PW, Harari AE, Getka EJ, Shakir KM. Combined levothyroxine plus liothyronine compared with levothyroxine alone in primary hypothyroidism: a randomized controlled trial. JAMA. 2003; 290:2952-2958.
QOL as measured by General Health Questionnaire (GHQ)-12 | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Besthesda, Maryland, United States

REFERENCES:
- [Derived] Shakir MKM, Brooks DI, McAninch EA, Fonseca TL, Mai VQ, Bianco AC, Hoang TD. Comparative Effectiveness of Levothyroxine, Desiccated Thyroid Extract, and Levothyroxine+Liothyronine in Hypothyroidism. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4400-e4413. doi: 10.1210/clinem/dgab478. PMID 34185829